CLINICAL TRIAL: NCT06410079
Title: Do Patients Under the Age of 50 Resume Equivalent Physical Activity Levels After Conventional Total Hip Replacement or Hip Resurfacing?
Brief Title: Difference in Return to Sports Activity After Hip Arthroplasty by THR or Resurfacing
Acronym: PTH-50
Status: Not yet recruiting | Type: Observational
Sponsor: Société Française de chirurgie de la Hanche et du Genou (Other)
Collaborators: Elsan (Other)
Responsible Party: Sponsor
Other Study IDs: 2023 A02666
Record Dates: First submitted 2024-05-03; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hip Arthrosis; Femur Head Necrosis
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- resurfacing: involves removing damaged cartilage and bone from the hip joint, half of the femoral head is cut, the neck and the other half are preserved, the acetabulum is covered by a metal cup
  Interventions: Procedure: total hip replacement
- total hip prosthesis: dual mobility total hip prosthesis in polyethylene, ceramic hip prosthesis, total hip prosthesis in ceramic or metal and polyethylene
  Interventions: Procedure: total hip replacement

INTERVENTIONS:
Procedure: total hip replacement — Replacement of the hip joint with a total prosthesis, a femoral stem, an acetabular cup, a joint head, in metal, ceramic, dual mobility or polyethylene

SUMMARY:
This study aims to evaluate the return to activity in younger patients under 50 years old after undergoing either total hip replacement (THR) or hip resurfacing, as performed in everyday practice. This research will be observational, meaning patients will not be randomly assigned to different treatment groups. To objectively assess participents; return to everyday, professional, and sports activities, validated questionnaires will be sent to participents in addition to routine clinical practice. The study will be prospective and comparative based on the type of prostheses used.

In order to capture the current practices of surgeons performing THR in participents under 50 years old in France, the study will be conducted at multiple centers across the country. Since hip resurfacing is performed only in certain centers, approximately half of the participating centers are experienced in this technique.

Participents typically resume activity between 3 and 6 months after THR. One year of post-operative follow-up allows for an accurate assessment of participents; recovery, unaffected by the surgery. Participents ; physical activity levels will be evaluated using the UCLA Activity Scale developed by surgeons to assess the activity levels of patients undergoing hip and arthroplasty.

DETAILED DESCRIPTION:
The literature is very scarce on Total Hip Arthroplasty(THA) in young patients. To date, there is no comparison on activity resumption based on prosthesis type on a national scale. Total Hip Arthrosplaty (THA) has been subject to a French registry since 2015 for patients operated by resurfacing , but no analysis of prosthesis wear has been conducted. A retrospective study with a follow-up exceeding 10 years is required to address this point and is the subject of another ongoing research. Resurfacing allows the preservation of anatomical elements but remains limited in France. The primary cause of THA revision identified is periprosthetic fracture. After resurfacing, a THA is performed, while after THA, only revision THA is possible but entails a longer operative time with a significant financial impact.

The aim of the research is to compare the level of physical activity at 1 year follow-up, according to the type of prostheses in adult patients under 50. It is part of presenting the practices of THA in young individuals in France during a symposium organized by the SFHG for 2025.

Research Hypothesis Regardless of the type of implants used, total hip arthroplasty yields excellent results in young patients with early resumption of activities, including sports. A meta-analysis of 11 studies comprising 2297 patients shows that 70%-90% of patients resumed sports activities within 6-12 months post-THA . A more recent systematic literature review confirms that 82% of patients have resumed sports activity on average at 6 months .

The research hypothesis is that there is no difference in physical activity at 1 year between patients operated with different types of prostheses, including dual mobility.

Justification of Methodological Choices Given the number of young patients undergoing THA per year in France , and considering a 5% margin of error and a 95% confidence interval, the sample size to be included is 500 patients.

A retrospective monocentric study is proposed given the scarcity of data in this young population. It will include adult patients under 50 operated on from 2015 to 2020. Participants will be divided into three groups according to the type of prosthesis: hip resurfacing, ;soft-hard THA, and hard-hard THA.

A comprehensive review of the medical records will be conducted to collect data.

Physical activity will be assessed at 1 year post-surgery using the International Physical Activity Questionnaire (IPAQ), a reliable and validated tool . The primary outcome is the level of physical activity at 1 year, and secondary outcomes include functional scores (HHS, WOMAC), complications, and prosthesis survival rate.

Ethical Considerations This study complies with the ethical principles outlined in the Declaration of Helsinki. Participant data will be anonymized to ensure confidentiality. Informed consent will be obtained from all participants.

Expected Results It is expected that there will be no significant difference in physical activity level at 1 year between patients operated with different types of prostheses. The results will provide valuable information on the optimal type of prosthesis for young patients undergoing THA and contribute to improving patient outcomes and satisfaction.

Primary objective The primary objective of the research is to compare the level of physical activity of participants at 1 year between those operated by resurfacing and those operated for a THA, taking into account their usual level.

Secondary objectives

The secondary objectives of the study are to:

1. Compare physical and professional activity:

* Compare the level of physical activity of patients at 1 year between the 4 studied prosthesis groups, taking into account their usual level.
* Compare the level of physical activity at 1 year to the preoperative level between the 2 groups and then between the 4 prosthesis groups.
* Compare the change in physical activity level between the 2 groups and then between the 4 prosthesis groups in relation to usual level and preoperative level
* Compare the time to return to physical and sporting activity in the year following hip arthroplasty.
* Compare the time to return to usual professional activity.
* Evaluate the quality of return to activity.
* Evaluate early complications after total hip arthroplasty.

  * Compare the participants postoperative experience.
  * Analyze the factors influencing the return to physical activity.
  * Describe the type of implant, surgical approach and clinical parameters in each group Evaluation criteria Main evaluation criterion The main evaluation criterion is the 1-year difference in the UCLA score measuring participants physical activity in relation to their usual level for the resurfacing group and for all THAs.

Secondary evaluation criteria

The secondary evaluation criteria corresponding to the secondary objectives are:

1. For each prosthesis group:

   * The 1-year difference in the UCLA score measuring the participants physical activity in relation to their usual level
   * The 1-year difference in the UCLA score measuring physical activity in relation to the preoperative level
   * The UCLA score at different times (usual level, preoperative, 6 weeks, 3 months, 6 months, 12 months).
   * The time to return to activities and sports
   * The time to return to usual professional activity
   * The quality of return to activity is evaluated by the Oxford hip functional scores.
   * Complications and the rate of revision surgery (if applicable) .Participants experience is measured by the SHV (Subjective Hip Value) Score and the Forgotten Hip Score (/100, 100=normal) at all study visits compared to the preoperative value.

     * The factors influencing the time to return to physical activity at the usual level in the year following prosthetic surgery taken into account for the analysis are patient-related parameters (rehabilitation or not, age, physical activity, medical history including inflammatory diseases), surgery-related parameters (type of implant, surgical approach and length of hospitalization)
     * The type of implant, surgical approach and clinical outcomes Research design Research scheme Observational, non-inferiority, non-randomized, prospective, multicenter, national study.

   Patients operated on the hip will be classified into 4 groups according to the type of prosthesis:
   * The resurfacing group
   * The THA group (hard-soft)
   * The THA group (dual mobility)
   * The THA group (hard-hard) Methods to limit bias Choice of centers Inclusion control Research Procedure The research procedure consists of collecting data from the medical records of patients followed in the context of current practice (demographics, anthropometry, comorbidities, medical history, etiology, surgery-related data, first mobilization, length of stay, discharge, type and duration of rehabilitation). In addition to current practice, patients will be asked to complete questionnaires on their return to activity (daily, professional and sports) with a systematic collection of postoperative events and any complications. No medical procedures or visits have been added in the context of this research.

   Questionnaires Assessing Physical Activity The patients; level of activity is assessed by the Devane score: it assesses work-related and/or sports activities. It is a score that gives an overall assessment of the participants level of activity or sedentary lifestyle rather than their actual sports practice. The score ranges from 1 to 5 depending on the participants answers, with 5 corresponding to the most intense activities .

   The participants pre-operative sports profile is assessed by 3 questions asked to the participant.

   Post-operative return to sports activity is assessed by 1 question (yes/no with 4 modalities to explain the reason for no). If the participant has resumed sports activity, 4 additional questions are asked about the frequency per week, whether it is the same activity, whether it is at the same level as before the intervention and the type of activity.

   The participant level of physical activity is assessed by the UCLA score, from the University of California, Los Angeles . This scale was originally developed by surgeons to assess the physical activity levels of patients who had undergone hip and knee arthroplasty . It is a 10-level, single-item scale, ranging from 10, for a patient who regularly participates in impact sports, to 1, for a patient who is completely inactive, dependent on others and unable to leave their home.

   Questionnaires Assessing Hip Function

   The functional results of the hip are assessed by the participant with the following questionnaires:

   . The Oxford Hip Score; (OHS-12 Delaunay et al, 2009) questionnaire is composed of 12 questions. It measures pain (on 6 items) and hip function (on 6 items) in relation to activities of daily living such as walking, the ability to dress, and sleep disturbances. Each question has 5 possible answers. Each corresponds to a value of 0 (= highest severity) to 4 (= total or almost total absence of symptoms). The sum of the answers to the questions is normalized on a scale between 0 and 100.

   The SHV (Subjective Hip Value) questionnaire is an analog evaluation scale coded from 0 to 100 (= Normal hip)

   The FJS (Forgotten Joint Score) HIP or Forgotten Hip Score is set at 100, with 100 corresponding to a normal hip .

   Other Questions Asked of the Patient Patients will be asked questions about bleeding, swelling, and wound healing in the days and weeks after surgery. Immediate complications and reoperation, if applicable, will be collected.

   In addition, patients will be asked about the duration of work stoppage and sports cessation before and after surgery.

   Treatments and Associated Procedures Authorized Associated Treatments/Procedures Any treatment necessary for the routine care of the participant is authorized.

   Prohibited Associated Treatments/Procedures No associated treatment or procedure is prohibited during the study.

   Conduct of the Research Research Schedule Duration of the inclusion period: 6 months Duration of participation for each participant: maximum 15 months Total duration of the research: 21 months

   Visit 1

   Visit 1 is the inclusion visit, corresponding to the pre-operative visit with the surgeon. It is conducted by the investigator physician and usually takes place between 3 and 1 month before the surgical procedure (D0). This visit includes:

   Providing the information sheet and explaining the research Verifying all eligibility criteria Obtaining the participants non-opposition by the physician Collecting demographic and anthropometric data (age, sex, height, weight) Collecting comorbidities and history of the hip and spine, etiology Visit 2

   Visit 2 corresponds to the sending of questionnaires by email to the participant 14 days before the surgical procedure D0 (Visit 3):

   Description of profession and activities (5 min) Degree of activity (Devane score) (1 min) Patients sport profile (1 min) Usual UCLA activity level and preoperative UCLA activity level (3 min) Self-questionnaires: Oxford questionnaire (20 min) Participant feelings by SHV and hip awareness FJS HIP (3 min) Collection of the duration of sports and professional cessation before surgery (2 min) A reminder for the primary endpoint is planned until the day before the procedure.

   Visit 3 Visit 3 corresponds to the hip surgery by resurfacing or total prosthesis placement according to the surgeons current practice.

   Surgical data will be collected such as the operated side, surgical approach, type of anesthesia, duration of the procedure, type of prosthesis and friction couple, surgical procedure and any immediate complications.

   Visit 4 Visit 4 corresponds to the collection of postoperative data from the participant during the postoperative period between the surgical procedure D0 (Visit 3) and the postoperative visit at 3 months (Visit 5).

   The following data will be collected during his/her hospital stay and then by email upon discharge:

   The first day of postoperative mobilization, discharge location, prescription of rehabilitation sessions Bleeding at D1 D3, D7 Edema at D21 and D42 Healing at D21 and D42 Participant feelings by the SHV at D28, D42, D70 UCLA physical activity level questionnaire at D42 Return to work at D28, D35, D42, D70 Surgical complications and any reoperation throughout follow-up Visit 5

   Visit 5 corresponds to the collection of data at the 3-month postoperative visit:

   Postoperative UCLA activity level Oxford questionnaire (sent 5 days before at D85-10min) Participants feelings SHV and hip awareness FJS Hip Edema Surgical complications and any reoperation Return to work and sports activities Collection of SAEs Visit 6

   Visit 6 corresponds to the collection of data at the 6-month postoperative visit:

   Postoperative UCLA activity level Oxford questionnaire (sent 5 days before Visit 6, at D175-10min) Participant feelings SHV and hip awareness FJS Hip Surgical complications and any reoperation Return to work and sports activities. End-of-Study Visit or Visit 7

   Visit 7 corresponds to the collection of data at the 12-month postoperative visit:

   Postoperative UCLA activity level Oxford questionnaire (sent 5 days before Visit 7, at D356-10min) Participant feelings SHV and hip awareness FJS Hip Surgical complications and any reoperation Return to work and sports activities, Postoperative duration of sports and professional cessation Collection of SAEs Study Termination Rules and Protocol Deviations Withdrawal, Consent Withdrawal and Lost to Follow-up A participant who no longer wishes to participate in this research, particularly in case of withdrawal or consent withdrawal, may do so at any time for any reason. He/she will no longer be followed up in the context of this protocol but will continue to receive the best possible care given his/her state of health and the current state of knowledge.

   Withdrawal is a decision by an included participant to exercise his/her right to discontinue his/her participation in a research study, at any time during the follow-up, without incurring any prejudice as a result and without having to justify himself/herself.

   Consent withdrawal is a decision by a participant to withdraw his/her participation in a research study and to exercise his/her right to revoke his/her informed consent, at any time during the follow-up and without incurring any prejudice as a result and without having to justify himself/herself.

   The investigator must assess whether it is possible to collect the variable on which the primary endpoint is based at the time of withdrawal/withdrawal. Withdrawals/withdrawals must be promptly notified to the coordinating investigator center, the sponsor and the data management and methodology center. The reasons, if known, and the date of withdrawal/withdrawal must be documented in the observation notebook and in the participants medical record.

   A participant is considered lost to follow-up when he/she stops the follow-up planned in the protocol for no reason known to the investigator, so that the data collection cannot be carried out as planned. In case of a lost-to-follow-up subject, the investigator will make every effort to get back in touch with the person.

   The observation notebook will be completed until the end of the study by documenting the reason for leaving.

   Research Termination Rules End of research or planned termination of research: end of participation of the last person who lends himself/herself to the research, also called last visit of the last participant included in the research.

   When the research has reached its planned term (planned termination), the end of the research must be declared to the ANSM and the CPP within 90 days.

   Early termination of research: the clinical research is stopped (definitively) in advance. This is the case, in particular, when the sponsor decides:

   Not to start the research despite the favorable opinion of a CPP Not to resume the research after having temporarily interrupted it or after its suspension by the ANSM.

   When the research is stopped (definitively) in advance, the end of the research must be declared to the ANSM within 15 days, indicating the reasons for this stop.

   Temporary suspension of research: the temporary suspension of a clinical research consists of:

   The cessation of the inclusion of new persons in this research. And/or the cessation of the administration of the tested product, if applicable, to all or part of the persons already included in the research.

   And/or the cessation of the acts provided for in the research protocol. Any decision by the sponsor to temporarily suspend the research must be immediately informed to the ANSM and the CPP concerned and, in a second step and within a maximum of 15 calendar days following the date of this suspension, a request for authorization for a substantial modification concerning this temporary suspension submitted to the ANSM and a request for an opinion to the CPP concerned.

   1.2.3. Premature Terminations The investigator may temporarily or permanently discontinue a participants contribution to the study for any reason that would best serve the participants interests, particularly in the event of an SAE. These participants will no longer be followed up in the context of this protocol but will continue to receive the best possible care given their state of health and current knowledge.

   The performance of a THP on the other side during the study or the occurrence of an SAE compromising the evaluation of the primary endpoint is a reason for premature termination.

   The study provides for early exit of participants who are in either of these situations. These participants will no longer be followed up in the context of this protocol but will continue to receive the best possible care given their state of health and current Premature Terminations The performance of a THP on the other side during the study or the occurrence of an SAE compromising the evaluation of the primary endpoint is a reason for premature termination.

   The study provides for early exit of participants who are in either of these situations. These participants will no longer be followed up in the context of this protocol but will continue to receive the best possible care given their state of health and current knowledge.

   For all premature study withdrawals, the investigator must document the reasons as completely as possible. The observation notebook will be completed until the end of the study.

   The study may be interrupted prematurely in the event of unexpected adverse events, SAEs, requiring a review of the medical strategies profile. Similarly, unforeseen events or new information relating to medical strategies may lead the sponsor to prematurely interrupt the study.

   Participants Included in Error A participant is considered to be included in error when he/she has actually been included in the research even though he/she did not meet all the eligibility criteria. Participants included in error must be discussed. They must continue to be followed up as planned by the protocol until a decision has been made by the sponsor in agreement with the study coordinating investigator.

   Protocol Deviations Deviations must be documented by the investigator. A protocol deviation may be discussed between the investigator and the sponsor. Even in the event of a protocol deviation, the participants follow-up must be conducted until the end of the protocol.

   Definitions Adverse Event (Article R.1123-46 of the Public Health Code) Any harmful manifestation occurring in a person who lends himself/herself to research involving the human person, whether or not this manifestation is related to the research or the product on which the research is carried out.

   Serious Adverse Event or Effect (Article R.1123-46 of the Public Health Code and ICH E2B Guide)

   Any adverse event that:

   Certain circumstances requiring hospitalization do not fall under the severity criterion of ;hospitalization such as:

   admission for social or administrative reasons, hospitalization predefined by the protocol, hospitalization for medical or surgical treatment scheduled before the research, day hospital stay. Adverse events likely to be related to a drug or product mentioned in Article R. 5121-150 to be declared to the Regional Pharmacovigilance Center (CRPV) on which it depends.

   Incidents or risks of incidents resulting from the use of a medical device to be reported to the local Matériovigilance correspondent.

   Monitoring and Reporting of Serious Adverse Events The study was non-interventional, no serious adverse events are expected related to this study.

ELIGIBILITY:
* Inclusion Criteria:
* Participant is male or female, aged 50 or under
* Participant is indicated for a primary THA or resurfacing procedure
* Participant agrees to complete and receive questionnaires by email
* Participant has been informed and has not objected to the collection and use of their data
* Exclusion Criteria:
* Participant is aged under 18 or over 50 years
* Participant has had a previous THA or resurfacing procedure
* Participant is scheduled for a THA on the other hip within the year
* Participant has severe physical and/or psychological health problems that, in the investigators opinion, may affect the participant's compliance with the study
* Participant is participating in another research study
* Participant is in the exclusion period of another research study that is still ongoing at the time of inclusion
* Participant is a protected person: an adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Participant is pregnant, breastfeeding or giving birth
* Participant is hospitalized without consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited by surgeons during orthopedic surgery consultations at each of the participating centers in the study. These consultations will take place between 3 and 1 month before the intervention. The purpose of the research will be explained to all patients who meet the eligibility criteria by the surgeon and an information sheet will be given to them. The physician will obtain the patients consent to participate in the research and their non-opposition to the collection and use of their data at least 14 days before the intervention, allowing sufficient time for the participant to reflect.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
UCLA hip score | Day 0, and 3 ,6,12 mounths
  The UCLA Hip Score is a validated measurement tool used to assess the level of physical activity in patients undergoing hip arthroplasty. It consists of a single-item scale ranging from 10 to 1. A score of 10 indicates regular participation in impact sports, while a score of 1 indicates complete inactivity and dependency on others. This score is utilized to evaluate the patient's functional outcome and activity level following hip surgery.

SECONDARY OUTCOMES:
Subjective Hip Value (SHV) Score | Days 14 and 3,6, 12 mounths
  evaluate patients' subjective perception of their hip function following hip surgery. It's typically assessed on a scale from 0 to 100, where 100 represents a fully functional, pain-free hip similar to its pre-surgery state. Patients rate their hip function based on their comfort, mobility, and overall satisfaction with the outcome of the surgery. This assessment provides valuable insight into the patient's experience and satisfaction with their hip replacement procedure
The Forgotten Joint Score (FJS) | Day 0, and 3 ,6,12 mounths
  It measures how "forgotten" the joint feels, with higher scores indicating that patients are less aware of the replaced joint during daily activities. The score typically ranges from 0 to 100, with 100 indicating that the joint feels completely forgotten or normal. This assessment provides valuable information on the patient's perception of their hip replacement and its impact on their quality of life
Oxford Hip Score (OHS) | Day 0, and 3 ,6,12 mounths
  12 questions used to assess the functional status and pain level of patients following hip replacement surgery. The questions cover activities of daily living such as walking, dressing, and sleeping, and patients rate their difficulty or pain level on a scale from 0 to 4 for each question. The total score ranges from 0 to 48, with lower scores indicating greater pain and functional limitation.
The DEVANE Score | Day 0, 12 mounths
  tool used to evaluate the level of activity or sedentariness in patients. It assesses both professional and recreational activities, providing an overall assessment of the patient's activity level rather than focusing solely on their athletic pursuits. The score ranges from 1 to 5 based on the patient's responses, with 5 indicating the most intense level of activity.
Age | Day 0
  Years
Gendre | Day 0
  Male, female
Implant type | Day 0
  implant type, resurfacing, dual mobility, ceramic, ceramic or polyethylene metal
Surgical approach | Day 0
  choice of surgical approach, anterior, posterior
Rehabilitation | 12 mounths
  rehabilitation, in a center, at home with a physiotherapist or without
medical and surgical history | Day 0
  nflammatory disease, polyarthritis, previous surgical procedures on the hip, spine

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Isida, MD, Principal Investigator — SFHG
Locations (1):
- Santé Atlantique, Saint-Herblain, Nantes, France

IPD SHARING:
Plan to Share IPD: No
the sponsor has not yet decided on the sharing, a meeting of all members of the association must take place soon to decide

REFERENCES:
- See also: official page of Société Française de chirurgie de la Hanche et du Genou — https://sfhg.fr/